CLINICAL TRIAL: NCT06574048
Title: Trial of Dexamethasone vs Placebo as an Adjunctive Therapy to Hyperbaric Oxygen Treatment HBO in Patients With Acute Carbon Monoxide Poisoning
Brief Title: Carbon Monoxide Hyperbaric Oxygen With Steroid Therapy
Acronym: COHOST
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0564-24-FB
Record Dates: First submitted 2024-08-22; First posted 2024-08-27 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Carbon Monoxide Poisoning; Carbon Monoxide Intoxication; Carbon Monoxide Encephalopathy; Carbon Monoxide-induced Parkinsonism
MeSH Terms: conditions — Carbon Monoxide Poisoning | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pharmacy will provide either saline or 10mg dexamethasone in saline in a masked fashion so that the clinical staff are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hyperbaric Oxygen Therapy with Dexamethasone (Experimental): Participants will be treated with hyperbaric oxygen (HBO) therapy within three days of acute carbon monoxide poisoning. Treatment is a minimum of three inpatient sessions. Participants will also receive 10 mg dexamethasone per day while receiving HBO therapy (minimum of two doses, maximum of five doses if participants' stay is longer than three days). After three treatment sessions, participants will discharge home, barring no other medical complications requiring further hospitalization. In addition, continued HBO therapy plus steroids will be offered if participants are still dealing with CO poisoning sequelae as determined by study outcome measures.
  Interventions: Drug: Dexamethasone
- Hyperbaric Oxygen Therapy with Placebo (Saline) (Placebo Comparator): Participants will be treated with hyperbaric oxygen (HBO) therapy within three days of acute carbon monoxide poisoning. Treatment is a minimum of three inpatient sessions. Participants will also a saline placebo instead of dexamethasone while receiving HBO therapy. After three treatment sessions, participants will discharge home, barring no other medical complications requiring further hospitalization. In addition, continued HBO therapy plus steroids will be offered if participants are still dealing with CO poisoning sequelae as determined by study outcome measures.
  Interventions: Drug: saline placebo

INTERVENTIONS:
Drug: saline placebo — IV saline bolus
  Other Names: nebulized normal saline (NS) placebo
  Arms: Hyperbaric Oxygen Therapy with Placebo (Saline)
Drug: Dexamethasone — 10mg IV Dexamethasone
  Other Names: Ozurdex, Maxidex, DexPak 10 day, DexPak 6 Day, LoCort, DoubleDex, ReadySharp dexamethasone, DexPak 13 Day, ZonaCort
  Arms: Hyperbaric Oxygen Therapy with Dexamethasone

SUMMARY:
Hyperbaric Oxygen Therapy (HBO) is routine treatment of carbon monoxide (CO) poisoning to prevent delayed neurological sequelae. This study looking to see if neurologic outcomes are improved with the addition of dexamethasone. CO poisoning can initiate a free radical mediated process that can instigate a demyelinating process resulting in long term neurological sequelae in some, but not all patients. In other demyelinating disorders, steroids are a part of first line treatment. HBO is already used for acute CO poisoning, so this pilot study will try to ascertain if the addition of steroids in concert with each hyperbaric oxygen session will yield improved outcomes.

DETAILED DESCRIPTION:
Hyperbaric Oxygen Therapy (HBO) is routine treatment of carbon monoxide (CO) poisoning to prevent delayed neurological sequelae. This study looking to see if neurologic outcomes are improved with the addition of dexamethasone. CO poisoning can initiate a free radical mediated process that can instigate a demyelinating process resulting in long term neurological sequelae in some, but not all patients. In other demyelinating disorders, steroids are a part of first line treatment. HBO is already used for acute CO poisoning, so this pilot study will try to ascertain if the addition of steroids in concert with each hyperbaric oxygen session will yield improved outcomes.

The control group will receive three HBO treatment sessions plus placebo. The treatment group will receive three HBO treatment sessions plus 10 mg Dexamethasone per day during HBO therapy (minimum of two doses, up to a maximum of five doses if participant stays for longer than three days). After three treatment sessions, the participant will be discharged home barring no other medical complications requiring further hospitalization. In two weeks, participants will return for follow-up testing and evaluation. Continued HBO therapy plus placebo as well as HBO therapy plus steroids for respective group members will be offered if participants are still dealing with CO poisoning sequelae as determined by our outcome measures. In addition, a 6 week and 12 week telephone follow-up will be conducted asking questions regarding memory, emotion, neurologic symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Acute CO poisoning, intentional or non-intentional exposure, receiving HBO treatment during hospitalization
* Age >18 years
* Nebraska Medicine admission

Exclusion Criteria:

* Mechanical ventilation
* No hospital admission or admission to hospital Critical Care Medicine Service
* Allergy to dexamethasone
* Pre-Existing neurological condition confounding outcome determination

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | Prior to hospital discharge after HBO therapy is no longer clinically warranted, and post-discharge at 2 weeks, 6 weeks, and 12 weeks.
  The Montreal Cognitive Assessment (MoCA) is a rapid screening instrument for mild cognitive dysfunction that assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuo-constructional skills, conceptual thinking, calculations, and orientation. The MoCA will be given in person while inpatient and via phone after discharge. Scored 0-30 Normal Cognitive performance 26 and above Mild impairment 18-25 Moderate impairment 10-17 Severe impairment 0-9

SECONDARY OUTCOMES:
Memory, Emotion, and Neurologic Symptoms | 6 weeks and 12 weeks post-treatment
  Post-treatment phone followup

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Cooper, MD, Principal Investigator — University of Nebraska
Locations (1):
- Nebraska Medicine, Hyperbaric Medicine Program, Clarkson Tower, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No